CLINICAL TRIAL: NCT03290378
Title: A Phase 3, Multicenter, Randomized, Double Blind, Three-Arm Study to Evaluate the Efficacy and Safety of Tramadol Infusion (AVE-901) Versus Placebo in the Management of Postoperative Pain Following Bunionectomy
Brief Title: Tramadol Versus Placebo in the Management of Postoperative Pain Following Bunionectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Avenue Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AVE-901-102
Record Dates: First submitted 2017-09-19; First posted 2017-09-21 (Actual); Results first posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2019-09

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia | interventions — Tramadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AVE-901 50 mg (Active Comparator)
  Interventions: Drug: Tramadol
- AVE-901 25 mg (Active Comparator)
  Interventions: Drug: Tramadol
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tramadol — IV; 25 mg or 50 mg, given at Hours 0, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, and 44
  Arms: AVE-901 25 mg; AVE-901 50 mg
Other: Placebo — IV; Placebo, given at Hours 0, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, and 44
  Arms: Placebo

SUMMARY:
The study evaluates the effectiveness and safety of IV tramadol compared to placebo managing postoperative pain following a bunionectomy

DETAILED DESCRIPTION:
(Non-clinical summary)

Tramadol is a centrally-acting synthetic analgesic of the aminocyclohexanol group with opioidlike effects. Tramadol is extensively metabolized following administration, which results in a number of enantiomeric metabolites that display different opioid-receptor binding properties, and monoaminergic reuptake inhibition.

ELIGIBILITY:
Key Inclusion Criteria:

* The patient is male or female 18-75 years of age undergoing unilateral first metatarsal bunionectomy surgery
* Willing to give consent and able to understand the study procedures
* Female patients must be of non-childbearing potential or be practicing a highly effective contraception
* The patient must be willing to be housed in a healthcare facility and able to receive parenteral analgesia for at least 72 hours after surgery.
* The patient meets definition of American Society of Anesthesiologists (ASA) Physical Class 1, or 2.

Exclusion Criteria:

* Patient is not expected to receive a continuous infusion nerve block as described in the Post-Op anesthetic procedures protocol
* Patient is undergoing bilateral or revision bunionectomy surgery
* The patient has allergy or hypersensitivity (or is intolerant) to opioids or tramadol The patient has known physical dependence on opioids
* The patient has taken other prior/concurrent chronic medications that have not been at a stable dose for at least 2 weeks prior to screening
* The patient is taking herbal or dietary supplements or medications that are moderate or strong inhibitors of CYP2D6 or CYP3A4 or inducers of CYP3A4
* The patient has taken monoamine oxidase (MAO) inhibitors, trazodone, or cyclobenzaprine within 14 days prior to surgery
* The patient cannot be withdrawn from medications (at least 7 days prior to surgery) that may lower the seizure threshold (e.g. anti-psychotic agents, MAOI inhibitors) or which increase serotonergic tone (e.g. selective serotonin reuptake inhibitors (SSRIs), serotonin norepinephrine reuptake inhibitors (SNRIs), tricyclic antidepressants, triptans).
* The patient has a history of epilepsy, or is known to be susceptible to seizures
* The patient has a history of Long QT Syndrome or a relative with this condition
* The patient has expressed suicidal ideation or is considered to be at risk of suicide.
* The patient is morbidly obese (body mass index [BMI] ≥ 40 kg/m2) or has documented sleep apnea requiring pharmacological or device intervention.
* Clinically significant abnormalities in the judgement of the Investigator
* The patient was administered an investigational product within 30 days prior to Screening.
* The patient has previously participated in a clinical study with AVE-901.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2018-04-11 (Actual); Study Completion 2018-04-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Trovare Clinical Research, Bakersfield, California
  - Lotus Clinical Research, Pasadena, California
  - Cheseapeake Research Group, LLC, Pasadena, Maryland
  - H.D. Research Corporation, Houston, Texas
  - Endeavor Clinical Trials, PA, San Antonio, Texas

REFERENCES:
- [Derived] Singla NK, Pollak R, Gottlieb I, Leiman D, Minkowitz H, Zimmerman J, Harnett M, Ryan M, Lu L, Reines S. Efficacy and Safety of Intravenously Administered Tramadol in Patients with Moderate to Severe Pain Following Bunionectomy: A Randomized, Double-Blind, Placebo-Controlled, Dose-Finding Study. Pain Ther. 2020 Dec;9(2):545-562. doi: 10.1007/s40122-020-00184-2. Epub 2020 Jul 18. PMID 32683644

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AVE-901 50 mg | AVE-901 25 mg | Placebo
Started | 140 | 133 | 136
Completed | 137 | 123 | 120
Not Completed | 3 | 10 | 16

BASELINE CHARACTERISTICS:
Population: Patient 03-042 was randomized to tramadol 25 mg but received tramadol 50 mg in error.
Groups:
- Total: Total of all reporting groups
Arm/Group | AVE-901 50 mg | AVE-901 25 mg | Placebo | Total
Number analyzed (Participants) | 139 | 134 | 136 | 409
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (13.51) | 44.5 (13.15) | 45.0 (13.44) | 45.2 (13.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 116 | 113 | 349
  Male | 19 | 18 | 23 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 51 | 46 | 52 | 149
  Not Hispanic or Latino | 88 | 88 | 84 | 260
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 4 | 7
  Asian | 2 | 3 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 29 | 38 | 37 | 104
  White | 104 | 88 | 88 | 280
  More than one race | 2 | 2 | 3 | 7
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 139 | 134 | 136 | 409
Previous opioid history [Count of Participants; unit: Participants]
  Yes | 42 | 52 | 47 | 141
  No | 97 | 82 | 89 | 268
American Society of Anesthesiology (ASA) Physical Classification [Count of Participants; unit: Participants] — Patient was to meet definition of American Society of Anesthesiologists (ASA) Physical Class of I or II:
  ASA I) normal healthy patient: healthy, non-smoking, no or minimal alcohol use) or
  ASA II) A patient with mild systemic disease: Mild diseases only without substantive functional limitations. Examples include (but not limited to): current smoker, social alcohol drinker, pregnancy, obesity (30<BMI<40), well-controlled DM/HTN, mild lug disease.
  Participants
    1 | 70 | 71 | 72 | 213
    2 | 69 | 63 | 64 | 196
Qualifying Categorical Pain Score [Count of Participants; unit: Participants] — The patient reported a score of moderate or severe on a 4-point categorical rating scale (with categories of none, mild, moderate, or severe)
  Participants
    Moderate | 89 | 80 | 75 | 244
    Severe | 50 | 54 | 61 | 165
BMI [Median (Standard Deviation); unit: kg/m2] — BMI Calculation: Sites used the NIH website BMI calculator: https://www.nhlbi.nih.gov/health/educational/lose_wt/BMI/bmicalc.htm
  kg/m2 | 27.9 (4.97) | 28.1 (5.48) | 28.3 (4.91) | 28.1 (5.12)
Qualifying Numerical Pain Rating Scale (NPRS) [Mean (Standard Deviation); unit: score on a scale] — Patient recorded a pain score ≥5, within 8 hours after removal of popliteal block, on an Numerical Pain Rating Scale (NPRS) where 0 is no pain and 10 is the worst pain imaginable. Patient needed to have a pain score of ≥5 to qualify for the study.
  Mean pain score per treatment group noted below.
  score on a scale | 6.7 (1.66) | 6.8 (1.39) | 6.9 (1.63) | 6.8 (1.56)

OUTCOME MEASURES:

1. Primary Outcome: The Sum of Pain Intensity Differences (SPID) Through 48 Hours Post First Dose
Description: Pain intensity was recorded using the Numerical Pain Rating Scale (NPRS) from 0 to 10, where 0 was no pain and 10 was the worst pain imaginable at hrs: .5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 34, 36, 38, 40, 42, 44, 46, 48. As higher pain scores indicate worse pain, a negative Pain Intensity Difference (PID) indicates less pain (improvement from baseline). Thus, SPID scores are expected to be negative if a patient's pain decreases over time, with the lower SPID values indicating greater reduction in pain intensity.
Time Frame: 48 hours post first dose
Population: One patient was randomized to tramadol 25 mg but received tramadol 50 mg in error.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | AVE-901 50 mg | AVE-901 25 mg | Placebo
Number analyzed (Participants) | 139 | 134 | 136
score on a scale | -122.8 [-135.14 to -110.50] | -110.9 [-123.64 to -98.17] | -97.8 [-110.60 to -85.00]
Statistical Analysis 1: Comparison: AVE-901 50 mg vs Placebo; Test type: Superiority; p < .005, ANCOVA

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | AVE-901 50 mg | AVE-901 25 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/140 | 0/133 | 0/136
Serious Adverse Events (participants affected / at risk) | 0/140 | 1/133 | 0/136
Other Adverse Events (participants affected / at risk) | 93/140 | 56/133 | 60/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AVE-901 50 mg (N=140) | AVE-901 25 mg (N=133) | Placebo (N=136)
non-cardiac chest pain (General disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AVE-901 50 mg (N=140) | AVE-901 25 mg (N=133) | Placebo (N=136)
Nausea (Gastrointestinal disorders) | 45 | 12 | 11
Headache (Nervous system disorders) | 8 | 14 | 13
Vomiting (Gastrointestinal disorders) | 28 | 4 | 5
Dizziness (Nervous system disorders) | 21 | 7 | 4
Infusion Site Pain (General disorders) | 11 | 5 | 10
Somnolence (Nervous system disorders) | 16 | 6 | 3
Infusion site extravasation (General disorders) | 5 | 7 | 5
Constipation (Gastrointestinal disorders) | 8 | 3 | 3
Pruritus generalized (Gastrointestinal disorders) | 4 | 3 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 3 | 2
Decreased Appetite (Gastrointestinal disorders) | 0 | 1 | 3
Muscle Twitching (Nervous system disorders) | 0 | 3 | 1
Rash (General disorders) | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/78/NCT03290378/Prot_SAP_000.pdf